CLINICAL TRIAL: NCT03511534
Title: Open/Aftercare Treatment for Participants Diagnosed With Obsessive Compulsive Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41165
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: OCD
Keywords: treatment, psychotherapy, pharmacotherapy
MeSH Terms: interventions — Psychotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Participants will choose to enter the psychotherapy or pharmacotherapy arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychotherapy (Active Comparator): Participants will receive evidenced based psychotherapy by a trained psychologist
  Interventions: Behavioral: Psychotherapy
- Pharmacotherapy (Active Comparator): Participants will receive pharmacotherapy by a psychiatrist
  Interventions: Other: Pharmacotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Evidenced based psychotherapy by a trained psychologist
  Arms: Psychotherapy
Other: Pharmacotherapy — Pharmacotherapy by a psychiatrist
  Arms: Pharmacotherapy

SUMMARY:
The purpose of this study is to provide participants diagnosed with obsessive compulsive disorder (OCD) and completed one of the active study protocols at the Rodriguez Lab, with open/aftercare treatment.

DETAILED DESCRIPTION:
After completing one of the active clinical studies participants have the option to enroll in this protocol that offers open treatment.

The goal is to compare two forms of current standard treatments, psychotherapy vs pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to speak and understand English
2. Capacity to consent (e.g. as determined by assessing the patient's understanding of the risks, benefits, and procedures of the study)
3. Completed an active study protocol at the Rodriguez Lab at Stanford University

Exclusion Criteria:

1. Children younger than 18
2. Active suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Up to 14 weeks
  Improvement in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Assistant Professor, Stanford University
Locations (1):
- Stanford University, Stanford, California, United States